CLINICAL TRIAL: NCT05090748
Title: A Pivotal Study for the Assessment of the Quality of Echocardiographic Clips When Obtained by Novice Users While Using the UltraSight Echocardiography Guidance (USEG) Software.
Brief Title: Study for the Assessment of the Quality of Echocardiographic Clips.
Status: Completed | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: USEG- 201
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Echocardiographic. — Echocardiographic test.

SUMMARY:
This study main objective is to evaluate the safety and efficacy of the UltraSight AI Guidance software. The investigational product is a software that guides the user to capture a high quality ultrasound image. The study will include healthcare professionals, not specialized in echocardiography, who will perform echocardiography by using UltraSight AI Guidance software, on subjects in the medical centers cardiac units.

DETAILED DESCRIPTION:
This pivotal study is a multi-center, multi-reader multi-case (MRMC) study, designed to assess the quality of the clips obtained by novice users when using the UltraSight AI Guidance software. Prior to the study start, there will be a pre-study training phase for training the novice users.

During the study, eligible subject will undergo the echocardiography examination twice on a single study visit (same day): once by one of the novice users when using the UltraSight AI Guidance software, and once by an expert sonographer without the aid of the software.

Each novice user will perform the examination on at least 20 subjects (with the aim that the number of examinations by each novice will be similar). All examinations will be sent to multiple Board certified cardiologists for their quality evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Subjects willing and able to give written informed consent.

Exclusion Criteria:

1. Emergency (non-elective) admission within 24 h prior to participating in the study
2. Female subjects who are pregnant (women of childbearing potential will perform a urine pregnancy test)
3. Unable to lie as required in all the classic positions for standard TTE exam: supine on back / left decubitus
4. Subjects who currently participate a clinical trial, involving interventional cardiac devices.
5. Subjects who have prior Echo exam with description of Low/Poor quality exam in the echo report
6. Subjects with BMI above 40
7. Subjects experiencing a known or suspected acute cardiac event
8. Subjects with severe chest wall deformity as per previous medical records and physical examination
9. Subjects who have undergone pneumonectomy
10. Subjects whose anatomy does not lend itself to yield diagnosable standard echocardiography clips (i.e. situs inversus with dextrocardia, single ventricle anatomy due to congenital heart disease, etc.).

    * A woman is of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis.).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male and female adults confirmed as eligible according to eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the echo examination sufficiency. | 1 year.
  The expert cardiologists will evaluate whether the echo examination quality obtained by novice users has sufficient to evaluate each of the primary endpoints:
  1. Sufficient quality to assess Left Ventricular (LV) size: (YES/NO)
  2. Sufficient quality to assess LV function: (Yes/No)
  3. Sufficient quality to assess Right Ventricular size: (Yes/No)
  4. Sufficient quality to assess presence of non-trivial pericardial effusion: (Yes/No)

SECONDARY OUTCOMES:
Evaluation of the echo examination quality. | 1 year.
  The expert cardiologists will evaluate whether the echo examination performed by novice users has sufficient quality to evaluate the following six (6) anatomic elements:
  1. Qualitative visual assessment of RV function: (Yes/No)
  2. Qualitative visual assessment of left atrium size: (Yes/No)
  3. Qualitative visual assessment of Aortic valve structure: (Yes/No)
  4. Qualitative visual assessment of Mitral valve structure: (Yes/No)
  5. Qualitative visual assessment of Tricuspid valve structure: (Yes/No)
  6. Qualitative visual assessment of IVC size: (Yes/No)
Evaluation of the echo examination diagnostic quality. | 1 year.
  The expert cardiologists will evaluate if each of the following 10 views taken by novice users can be considered of diagnostic quality:
  * Apical 4 chamber
  * Apical 2 chamber
  * Apical 3 chamber
  * Apical 5 chamber
  * Para Sternal Long Axis
  * Para Sternal short axis - Aortic Valve (AV)
  * Para Sternal short axis - Mitral Valve (MV)
  * Para Sternal short axis - Papillary Muscle (PM)
  * Sub Costal - 4 chamber
  * Sub Costal - Inferior Vena Cava (IVC) In order to assess intra-cardiologist variability, a repeated assessment of the expert cardiologist analysis will be done in 10% of the exams.

OTHER OUTCOMES:
Safety outcome. | 1 year.
  Adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lang, MD, Principal Investigator — U of Chicago; Federico Asch, MD, Principal Investigator — Medstar Health Research Institute; Praveen Mehrotra, MD, Principal Investigator — Thomas Jefferson University; Bijoy Khandheria, MD, Principal Investigator — Aurora Saint Luke Medical Center; Robert Klampfner, MD, Principal Investigator — Sheba Medical Center; Danny Spigelstein, MD, Study Director — UltraSight
Locations (3):
- United States (2):
  - University of Chicago Medicine, Chicago, Illinois
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Sheba MC, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No